CLINICAL TRIAL: NCT05244408
Title: "SCRIBBLE" Spinal Cord Injury Blood Biomarker Longitudinal Evaluation
Acronym: SCRIBBLE
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Brian Kwon, Principal Investigator, University of British Columbia
Other Study IDs: H22-00258
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Acute Spinal Cord Injury; Acute Spinal Paralysis; Spinal Cord Injuries; Trauma, Spinal Cord
Keywords: Serum; Biomarkers
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCI Subjects: Patients who suffer a traumatic spinal cord injury who meet the following inclusion criteria are eligible for admission into the study as "SCI subjects":
- Non-SCI Spine Trauma Control Subjects.: Patients who suffer a fracture or dislocation of their spinal column but without neurologic injury are eligible for admission into the study as "Non-SCI Spine Trauma Control Subjects"

SUMMARY:
Prospective, single center study designed to assess blood biomarkers for classifying injury severity and predict neurologic recovery in traumatic spinal cord injured (SCI) patients.

Study will also establish the accuracy of point to care devices for SCI blood biomarkers and support the biospecimen collection for the International Spinal Cord Injury Biobank (ISCIB).

DETAILED DESCRIPTION:
This single center study at Vancouver General Hospital (VGH) will enroll patients with acute traumatic cervical and thoracic SCI who will have blood samples obtained daily for the first week post-injury. They will then have follow-up neurologic assessments at 6 and 12 months post-injury. The specific aims of the study are to:

1. Validate serum Neurofilament Light Chain (NF-L) and Glial Fibrillary Acidic Protein (GFAP) as biomarkers of acute SCI for classifying injury severity and predicting neurologic recovery.
2. Establish the relationship between serum and plasma levels of NF-L and GFAP.
3. Establish the accuracy of point-of-care devices for measuring GFAP.
4. Support biospecimen collection for the International Spinal Cord Injury Biobank (ISCIB).

ELIGIBILITY:
Inclusion Criteria

SCI Participants. Patients who suffer a traumatic spinal cord injury who meet the following inclusion criteria are eligible for admission into the study as "SCI participants":

* Male or Female ≥ 19 years of age
* Blunt (non-penetrating) traumatic spinal cord injury
* Baseline neurologic impairment deemed "complete"(AIS A) or "incomplete" (AIS B, C, D)
* Bony spinal level involvement between C0 and L1 inclusive
* Ability to have initial blood sample drawn within 24 hours of injury
* Have either an arterial line, central line, or intravenous line for collecting blood samples
* Able and willing to provide informed consent

Non-SCI Spine Trauma Control Participants. Patients who suffer a fracture or dislocation of their spinal column without neurologic injury who meet the following inclusion criteria are eligible for admission into the study as "Non-SCI Spine Trauma Control Participants":

* Male or Female ≥ 19 years of age
* Traumatic spinal fracture between C0 and L1 without spinal cord injury
* Collection of initial blood sample within 24 hours of injury
* Have either an arterial line, central line, or intravenous line for collecting blood samples
* Able and willing to provide informed consent

Exclusion Criteria

Patients who fulfill any of the following criteria are not eligible for admission into the study:

* Penetrating spinal cord injury (e.g. gunshot, stab)
* Spinal cord injury with sensory deficit only (i.e. no motor deficit)
* Spinal injury below L1
* Isolated radiculopathy without fracture
* Isolated cauda equina injury
* Pre-existing thromboembolic disease or coagulopathy (disorders related to blood clotting), such as haemophilia or von Willebrand's disease
* Have any other medical condition that in the investigator's opinion would render the study procedures dangerous or impair their ability to receive treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants for this study will be recruited at Vancouver General Hospital. The study will include two groups/cohorts:
  SCI Subjects. Patients who suffer a traumatic spinal cord injury who meet the following inclusion criteria are eligible for admission into the study as "SCI subjects":
  Non-SCI Spine Trauma Control Subjects. Patients who suffer a fracture or dislocation of their spinal column but without neurologic injury are eligible for admission into the study as "Non-SCI Spine Trauma Control Subjects" if they meet the following inclusion criteria:
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Levels of specific biochemical markers in blood | Day 1 - 7
  Daily serum samples will be collected to assess serum GFAP and NF-L as biomarkers of acute SCI for classifying injury severity and predicting neurologic recovery

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examination | 12 Months
  Neurologic recovery over time will be measured using the ISNCSCI examination - at Baseline, Month 6 and Month 12. Our outcome measure will be the change in total motor score at 6 months post-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kwon, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada